CLINICAL TRIAL: NCT02564939
Title: Randomized, Double Blind, Placebo-Controlled Clinical Trial Evaluating Ramelteon in the Prevention of Delirium
Brief Title: Ramelteon Prevention of Delirium - RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Robert Dicks, Director Geriatrics, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HHC-2015-0073
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Delirium
Keywords: prevention
MeSH Terms: conditions — Delirium | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ramelteon (Active Comparator): receive ramelteon
  Interventions: Drug: ramelteon
- placebo (Placebo Comparator): receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ramelteon — double-blind RCT
  Other Names: Rozerem
  Arms: ramelteon
Drug: Placebo — double-blind RCT
  Arms: placebo

SUMMARY:
Delirium is a common morbid condition in hospitalized adults. Treatment of delirium has been unsatisfactory and prevention is the preferred goal. Based on limited experimental research, ramelteon appears to have promise for prevention. This study will evaluate ramelteon in prevention of delirium in a hospitalized adult population age 65+ in a double-blinded RCT.

DETAILED DESCRIPTION:
Delirium is a very common condition that is associated with significant complications in hospitalized adults.

The manifestations of delirium are the result of a disturbance of brain functioning, the causes of which include a very wide array of illnesses, intoxications, and stresses. Delirium has been estimated to affect 20-50% of hospitalized patients, and to be associated with longer hospital stay (2x), greater likelihood of discharge to nursing home (2x), and higher rate of death (2x). 20% have delirium on admission. Patients who experience delirium may have persistent confusion (cognitive impairment). In 20%, this confusion appears to be permanent. Treatment of delirium has been unsatisfactory. Once it develops, no therapy or intervention has demonstrated a meaningful reduction of delirium associated complications. Prevention is clearly the preferred goal. Based on limited reports, ramelteon appears to have the most promise for prevention. Ramelteon, FDA approved (2005) as a nonscheduled prescription hypnotic agent, is generally considered safe and effective with no serious associated side effects, and no limitation of duration of use. It is related to melatonin in action and shares sleep promoting effects (reduced sleep latency) and improvement in coordination of circadian cycles. A recent randomized placebo-controlled single blinded trial of ramelteon treated 33 patients with ramelteon 8 mg/d. The researchers reported that ramelteon was associated with a dramatically lower risk of delirium (3% vs 32%; P = .003), with a relative risk of 0.09. Estimates of time to develop delirium were delayed for ramelteon compared to placebo, and the frequency of delirium was significantly lower in ramelteon compared to placebo (P = .002). There were significant limitations of this study, however, including a very high exclusion rate (1059 of 1126 [94%] patients assessed were excluded), a 24+ hour delay in initiation of study agent, a small sample size, and unclear sampling bias. The investigators propose a clinical trial of ramelteon to prevent delirium in patients admitted to Hartford Hospital. Hartford Hospital is in a unique position to conduct this study having established the ADAPT program to systematically apply best practices to the assessment and management of delirium. A registry of patients screened contains all of the screening results (over 1.5 million CAM screens on nearly 91,000 patients). Our study will permit us to evaluate the recent limited research findings regarding ramelteon in a larger general adult hospitalized population, and evaluate the potential benefit of treatment started earlier in the course of a hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* from designated nursing units

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
delirium | through study completion, anticipate completion at 1 year
  delirium as determined by CAM screening and expert review

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Dicks, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States